CLINICAL TRIAL: NCT00000807
Title: Phase II Evaluation of Low-Dose Oral Etoposide for the Treatment of Relapsed or Progressed AIDS-Related Kaposi's Sarcoma After Systemic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 269; 11245 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Sarcoma, Kaposi; Etoposide; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Etoposide

INTERVENTIONS:
Drug: Etoposide

SUMMARY:
To assess the toxicity, tumor response rate, and effect on quality of life of daily low-dose etoposide administered for 7 consecutive days every other week in patients with AIDS-related Kaposi's sarcoma that has relapsed or progressed after systemic chemotherapy.

Etoposide may be at least as, or even more, effective and less myelotoxic when given in low doses over prolonged periods of time.

DETAILED DESCRIPTION:
Etoposide may be at least as, or even more, effective and less myelotoxic when given in low doses over prolonged periods of time.

Patients receive low-dose oral etoposide on days 1 through 7 of every 2-week cycle. Patients who achieve a complete or partial response after two cycles and have no toxicity greater than grade 2 may have their dose escalated for subsequent cycles. If there are no responses to therapy among the first 14 evaluable patients, the study will close; if there is at least one objective response to therapy among the first 14 evaluable patients, enrollment will continue until all 41 patients are enrolled. Patients continue therapy until maximal tumor response (either stable disease or complete response) is achieved or disease progression occurs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Maintenance therapy for opportunistic infections.

Patients must have:

* HIV infection.
* Kaposi's sarcoma that has relapsed or progressed.
* Mucocutaneous lesions (15 or more) and/or symptomatic mucosal lesions and/or visceral Kaposi's sarcoma (symptomatic lymphedema qualifies patients in the absence of these three conditions).
* NO active acute opportunistic infections requiring treatment with myelosuppressive antibiotics (maintenance for OIs is permitted).
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* This study is approved for prisoner participation.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Other active malignancies except basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Grade 3 or worse peripheral neuropathy.
* Altered mental status that would prevent informed consent or prevent study compliance.

Patients with the following prior condition are excluded:

Neuropsychiatric history.

Prior Medication:

Excluded:

* Prior etoposide.
* Any other anti-KS drugs within 14 days prior to study entry.
* Any investigational drug other than antiretrovirals within 14 days prior to study entry.
* Any prior investigational agent, if given as the ONLY prior treatment for KS.

Prior Treatment:

Excluded:

* Radiation therapy within 7 days prior to study entry.

Continued alcohol consumption or continued intravenous drug use that would impair ability to comply with study requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41
Dates: Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Von Roenn JH, Study Chair; Paredes J, Study Chair
Locations (20):
- United States (20):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - K Norris Cancer Hosp / Los Angeles County - USC Med Ctr, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Denver Dept of Health and Hosps, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Yale Univ / New Haven, New Haven, Connecticut
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Boston Med Ctr, Boston, Massachusetts
  - Adirondack Med Ctr at Saranac Lake, Albany, New York
  - Albany Med College / Division of HIV Medicine A158, Albany, New York
  - Mid - Hudson Care Ctr, Albany, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Saint Clare's Hosp and Health Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Mans D, Sprinz E, Sander I, Kalakun F, Jung G, Prolla G, Schwartsmann G. A phase II study of oral etoposide (VP-16) in AIDS-related Kaposi's sarcoma (KS). Int Conf AIDS. 1994 Aug 7-12;10(1):173 (abstract no PB0118)
- [Background] Evans SR, Krown SE, Testa MA, Cooley TP, Von Roenn JH. Phase II evaluation of low-dose oral etoposide for the treatment of relapsed or progressive AIDS-related Kaposi's sarcoma: an AIDS Clinical Trials Group clinical study. J Clin Oncol. 2002 Aug 1;20(15):3236-41. doi: 10.1200/JCO.2002.12.038. PMID 12149296